CLINICAL TRIAL: NCT06847516
Title: Predictors of Clinical and Neurological Outcome in Traumatic Posterior Fossa Epidural Hematoma
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Helal sayed ali, residant doctor, Assiut University
Other Study IDs: clinical +NeurologicalPFEH
Record Dates: First submitted 2025-02-21; First posted 2025-02-26 (Actual); Last update posted 2025-02-26 (Actual); Status verified 2025-02

CONDITIONS: Posterior Fossa Epidural Hematoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Group A: patients admitted to Neurosurgery department withTraumatic Posterior fossa epidural hematoma

SUMMARY:
The posterior fossa is a small space in the skull containing the brainstem and cerebellum. If a mass such as a hemorrhage grows in this region, particularly the brainstem and 4th ventricle, it can block the normal flow of cerebral spinal fluid leading to hydrocephalus, increased intracranial pressure.Posterior fossa extradural hematoma (PFEDH) is a rare neurosurgical entity, resulting in rapid clinical deterioration. The accumulation of blood in a potentially small space between the dura and occipital bone cause compression of the brain stem.These hematomas constitute almost 4% to 12.9% of all extradural hematoma cases.

The extradural hematomas of the posterior fossa may be categorized as acute or delayed defined with respect to the brainstem compression appearing within or after 24 hours of injury, respectively. Acute PFEDH is characterized by medullar failure, occipital trauma associated with severe pain in the nuchal area, altered consciousness followed by rapid brainstem compression, respiratory depression, and subsequent death if not treated timely and appropriately.Whereas, headache, neck pain, dysfunction of lower cranial nerve in response to PF lesions and cerebellar signs. The clinical features of PFEDH are nonspecific; it may include occipital headache, vomiting due to raised intracranial pressure, and decreased consciousness level leading to death. The skull fractures must be considered as a predisposing factor for the development of delayed extradural hematomas.

The aim of this study is :

* To evaluate the outcome of patients with traumatic post fossa Epidural hematoma
* list the predictors of outcome for patients with post fossa Epidural hematoma

ELIGIBILITY:
Inclusion Criteria:

* Any age
* Traumatic Posterior fossa epidural hematoma

Exclusion Criteria:

* Spontaneous type of epidural heamatoma

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: patients with Traumatic Posterior fossa epidural hematoma
Sampling Method: Probability Sample
Enrollment: 94 (Estimated)
Dates: Start 2025-03-01 (Estimated); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-05-01 (Estimated)

PRIMARY OUTCOMES:
The postoperative GOS score | 30 day
  he Glasgow outcome scale (GOS). GOS score four and five were considered good recovery outcomes, GOS 2 and 3 indicated poor outcomes, and OS one indicated mortality.